CLINICAL TRIAL: NCT06695767
Title: Neurobehavioral Therapy For Epilepsy And Major Depressive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Melissa Fadipe, Student, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-53437
Record Dates: First submitted 2024-11-09; First posted 2024-11-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Epilepsy
Keywords: veterans
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurobehavioral therapy (Experimental)
  Interventions: Behavioral: Neurobehavioral therapy

INTERVENTIONS:
Behavioral: Neurobehavioral therapy — Participants will receive an introduction session and 12 1-hour long online sessions once per week for a total of 12 weeks that are guided by the investigator who is trained in NBT.Participants will engage in tools to aid in assuming control over their seizures; contextualize their environment; identify moods, situations, and thoughts; train healthy communication and support seeking; understand central nervous system medications and seizures; conduct a functional behavioral analysis; learn relaxation techniques; examine external stressors and internal triggers; and prepare for life after the intervention. Participants will be asked to complete weekly homework, thought records, seizure logs that are found in their workbooks and to engage in journal entries.

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of an online group Neuro-behavioral Therapy (NBT) with text messaging intervention for Veterans with epilepsy and major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* English speaking veterans
* has home internet access
* has access to and familiarity in using a computer or tablet at least weekly
* Asymptomatic patients with chronic conditions
* has access to a mobile device with Short Message Service (SMS) text and picture capability
* has an active clinical diagnosis of major depressive disorder based on the International Classification of Diseases, 10th version (ICD-10)
* has an ICD-10 diagnosis of epilepsy with at least one seizure documented within the last five years

Exclusion Criteria:

* pregnancy
* Veterans that have current suicidal ideation
* have active psychosis; and have an ICD-10 diagnosis of psychogenic non-epileptic seizures or conversion disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-02-06 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | post intervention (14 weeks after baseline)
  This is defined as the number enrolled divided by the number of eligible participants screened
Retention rate | post intervention (14 weeks after baseline)
  This is defined as the number completing the study/number enrolled at baseline
Session attendance rate (proportion of sessions attended) | post intervention (14 weeks after baseline)
Homework completion rate (proportion of homework assignments completed) | post intervention (14 weeks after baseline)
User satisfaction as assessed by The Participant Satisfaction Survey | post intervention (14 weeks after baseline)
  This is a 16 item questionnaire and the first 10 questions are scored from 1( strongly disagree)to 5(strongly agree) for a maximum score of 50, higher score indicating better outcome

SECONDARY OUTCOMES:
Change in depression as assessed by the Patient Health Questionnaire-9 (PHQ-9), | baseline, end of session 12 (12 weeks form baseline)
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(Nearly every day), for a score range of 1-27, higher score indicating worse outcome
Change in quality of Life as assessed by the Quality of Life in Epilepsy Inventory-10 (QOLIE-10) | baseline, end of session 12(12 weeks form baseline)
  This is a 10 item questionnaire , with scores ranging from 0-100, with a higher score indicating better quality of life.
Change resilience as assessed by the Connor-Davidson Resilience Scale (CD-RISC) | baseline, end of session 12(12 weeks form baseline)
  This is a 25 item questionnaire, each rated on a 5-point scale from 0(not true at all) to 4(true nearly all the time), with higher scores reflecting greater resilience.
Change in efficacy in the self management of epilepsy as assessed by the Epilepsy Self-Efficacy Scale (ESES) | baseline, end of session 12(12 weeks form baseline)
  This is a 33 item questionnaire , rated on a 11-point Likert scale, ranging from 0(I cannot do it at all) to 10(sure I can do) for a maximum score of 330, higher score indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Fadipe, MSN, APRN, FNP-C, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The University of Texas health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No